CLINICAL TRIAL: NCT07358923
Title: Accuracy of Modified Milan Ultrasound Criteria in Assessing Disease Activity and Severity in Moderate-to-Severe Ulcerative Colitis: a Pilot Study
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mariangela Allocca, MD, PhD, IRCCS San Raffaele
Other Study IDs: Modified MUC
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Colon biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Longitudinal prospective monocentric observational study in which patients to start Mirikizumab for normal clinical practice will be followed for 24 weeks. Based on the findings in the comparison between US (IUS and TPUS) and endoscopy, the study aim is to build up a modified MUC (Milan Ultrasound Criteria) scoring system taking each colonic segment and the rectum into account, developing non-invasive quantitative ultrasound-based criteria to identify patients with active UC and assess its severity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of UC according to ECCO guidelines
* Patients with active moderate-to-severe disease defined as MES

  ≥ 2
* Patients undergoing advanced therapies with mirikizumab according to clinical judgement
* Patients who provide written informed consent

Exclusion Criteria:

* Age < 18 years
* Patients with unclassified colitis or other gastrointestinal conditions
* Patients with current infections or other severe comorbidity, including liver, kidney or cardiac failure, which contraindicate the initiation of advanced therapy
* Patients unable or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is a population of adult patients with confirmed diagnosis of UC according to ECCO guidelines with an active moderate-to-severe disease defined as MES ≥ 2 and who have indication to undergo advanced therapies with mirikizumab according to clinical judgement
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
To prospectively compare the diagnostic accuracy of modified MUC versus endoscopy (reference standard), in assessing disease activity and severity in UC. | IUS, TPUS and endoscopy will be performed at baseline and at week 24 (±2).